CLINICAL TRIAL: NCT00314600
Title: Above Elbow Cast in Non-Dislocated Both-Bone Midshaft Forearm Fractures in Children: Necessity or Needless Cruelty? A Randomized Trial
Brief Title: Treatment of Non-Dislocated Midshaft Both-Bone Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colaris, Joost, M.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Colaris02
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2007-02-26 (Estimated); Status verified 2006-11

CONDITIONS: Fracture
Keywords: Fracture; Forearm; Midshaft; Child; Cast
MeSH Terms: conditions — Fractures, Bone

INTERVENTIONS:
Device: above and below elbow cast

SUMMARY:
The investigators created a randomized clinical trial to find out what kind of treatment is optimal for non-dislocated both-bone midshaft forearm fractures.

DETAILED DESCRIPTION:
Children who arrive at the emergency unit with a non-dislocated both-bone midshaft forearm fracture will be asked to join the trial. After informed consent we will do a randomization between 6 weeks above elbow cast and 3 weeks above elbow cast in combination with 3 weeks under elbow cast.

Outpatient clinic visits till a follow-up of 6 months. During these visits we will investigate: consolidation and dislocation on X-ray, function of both arms, complaints in daily living and complications.

ELIGIBILITY:
Inclusion Criteria:

* Both-bone midshaft forearm fracture
* Age < 16 years old

Exclusion Criteria:

* Dislocation
* Fracture older than 1 week
* No informed consent
* Refracture
* Open fracture (Gustillo 2 and 3)
* Torus fractures of both ulna and radius

Max Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60
Dates: Start 2006-01

PRIMARY OUTCOMES:
pronation and supination

SECONDARY OUTCOMES:
complications, function, esthetics, complaints in daily living, X-rays

CONTACTS AND LOCATIONS:
Overall Officials: Joost W Colaris, M.D., Principal Investigator — HAGA/Erasmus Medical Centre
Locations (2):
- Netherlands (2):
  - Erasmus Medical Centre, Sophia Children's Hospital, Rotterdam, South Holland
  - HAGA, Juliana Children's Hospital, The Hague, South Holland

REFERENCES:
- [Derived] Colaris JW, Reijman M, Allema JH, Biter LU, Bloem RM, van de Ven CP, de Vries MR, Kerver AJ, Verhaar JA. Early conversion to below-elbow cast for non-reduced diaphyseal both-bone forearm fractures in children is safe: preliminary results of a multicentre randomised controlled trial. Arch Orthop Trauma Surg. 2013 Oct;133(10):1407-14. doi: 10.1007/s00402-013-1812-8. Epub 2013 Jul 17. PMID 23860674